CLINICAL TRIAL: NCT07017803
Title: Molecular Epidemiology, Strains Genotyping of Multi-drug Resistant Tuberculosis Circulating in Central Africa Region
Acronym: MESTCAR
Status: Not yet recruiting | Type: Observational
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: Fondation Congolaise pour la Recherche Médicale (Unknown); Centre Pasteur du Cameroun (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: CEI-004/2025
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis, Multi Drug Resistant; Strains; Molecular Epidemiology; Multi Drug Resistant Tuberculosis; Central Africa
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Multidrug-resistant tuberculosis (MDR-TB) poses a significant challenge in Central Africa. Understanding the molecular epidemiology and genotypic characteristics of MDR-TB strains is crucial for effective control measures. This is highlighted by the emergence of mutations encoding resistance to bed aquiline and quinolones which may impact the roll out of the newly recommended Bedaquiline, Pretomanid, Linezolid and Moxifloxacin (BPaLM) regimens.

It is also worth noting that there is increasing evidence of the significance of TB lineage in the outcome of infection, the approach in the study will provide both information on chains of transmission and lineage.

ELIGIBILITY:
Inclusion Criteria:

* All GeneXpert positive TB patients and participants who provide written informed consent will be screened for the study. Participants aged above 8 who can provide sputum will also be screened.
* Patients enrolled in the tuberculosis epidemiology (TB-EPI) study and eligible for MESTCAR will be enrolled without any additional consent form as the data to be collected for the two studies will be shared and no additional process is needed.

Exclusion Criteria:

* Samples which do not meet the quality criteria.

  * Samples not enough to perform all of the laboratory process
  * Samples contaminated

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be all TB presumptive patients who will be diagnosed and willing to participate in the selected facilities in the three countries, the different sites involved in the study are Institut Pasteur de Yaoundé (Cameroon), Centre de Recherche Medicales de Lambaréné (Gabon) and Laboratoire National de Reference de Tuberculose du Congo (Republic of Congo). In Gabon, this study will be included in the ongoing sequencing TB studys. Samples collected for ongoing TB study will be used to avoid competing sample collection. Two or more separate aliquot storage samples will be used for METSCAR and TB-EPI studies. This, together with the fact that the workgroups overlap 100%, will allow the ongoing studies in the group to be performed complementarily.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of drug-resistant strains with characterised resistance mutations | 6 months
Proportion of strains with new/undefined mutations among those with unexplained phenotypic resistance | 6 months
Proportion of cases demonstrating transmission links, overall and between countries | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ayôla Akim ADEGNIKA, Study Director — Centre de Recherches Medicales de Lambarene